CLINICAL TRIAL: NCT00793559
Title: Terlipressin Administration in Septic Shock Refractory to Catecholamines Bolus vs. Continuous Drip-Phase II
Brief Title: Terlipressin Administration in Septic Shock Refractory to Catecholamines
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr Yuval Leonov, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 161/08
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Septic Shock
Keywords: septic shock refractory to catecholamines
MeSH Terms: conditions — Shock, Septic | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- terlipressin bolus (Active Comparator): 1 mg of terlipressin received one time only
  Interventions: Drug: terlipressin
- terlipressin drip (Experimental)
  Interventions: Drug: terlipressin

INTERVENTIONS:
Drug: terlipressin — 1 mg of terlipressin one time only
  Other Names: glypressin
  Arms: terlipressin bolus
Drug: terlipressin — 1 mg of terlipressin in 50 cc of NS given at a drip of a total of 6 h
  Arms: terlipressin drip

SUMMARY:
terlipressin is given to refractory septic shock patients who do not respond to noradrenalin in Israel and Europe. It is given by bolus injection. we attempt to investigate weather it is better to give it by continuous drip and avoid abrupt changes in BP and heart function

ELIGIBILITY:
Inclusion Criteria:

* septic shock patients receiving above 0.5 mcg/kg NA

Exclusion Criteria:

* allergy to terlipressin, CHF, IHD, pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
CI, SVR,HR,BP, noradrenalin administration,renal function | 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Tal Mann, Dr, Study Director — Asaf Harofeh
Locations (1):
- Asaf Harofeh MC, Zrifin, Israel